CLINICAL TRIAL: NCT04325438
Title: The Impact of Pharmacists' Interventions on the Quality of Life of HIV-TB Co-infection Outpatients in Indonesia: a Therapeutic Drug Monitoring (TDM) Approach
Brief Title: The Impact of Pharmacists' Interventions on the Quality of Life of HIV-TB Co-infection Outpatients in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bekasi City Public Hospital (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Principal Investigator, Lusiana Rusdi Idrus, Pharmacist, Bekasi City Public Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HIVTB-INDO2017
Record Dates: First submitted 2019-08-01; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Pharmaceutical Care; HIV/AIDS; Tuberculosis
Keywords: Pharmaceutical care; Pharmacists' interventions; human immunodeficiency virus; tuberculosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis | interventions — Pharmaceutical Services

STUDY DESIGN:
Intervention Model Description: Stepped wedge design trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmaceutical Care (Experimental): Groups with usual care by health professionals and additional health interventions provided by pharmacists. Number of intervention groups in each cluster is different, depending on the starting time of the intervention.
  Interventions: Other: Pharmaceutical Care
- Non-Pharmaceutical Care (No Intervention): Groups with usual care from health providers other than pharmacists. Number of intervention groups in each cluster is different, depending on the starting time of the intervention.

INTERVENTIONS:
Other: Pharmaceutical Care — Pharmaceutical care interventions are categorised into 2 aspects:
  1. Pharmacists' expertise aspect: medications review, identification and solution for the drug-related problem, adverse events, and other medication-related clinical problems. Therapeutic drug monitoring (TDM) is performed for any dose adjustment to the Rifampicin.
  2. Motivational behavioral intervention to improve medication adherence (i.e. medications information and counseling to study participants).
  Arms: Pharmaceutical Care

SUMMARY:
Rationale:

The co-infection of human immunodeficiency virus (HIV) and tuberculosis (TB) diseases presents further problems to patient's adherence due to high pill burden and adverse effects in the drug combination therapy. This situation is also a risk of the increase of multi-drug resistant TB and may affect the quality of life of patients. However, the prevalence of non-adherence has not been studied much in these patients in Indonesia, especially in West Java with several HIV patients who are still struggling with TB as their opportunistic infection. Pharmacist interventions in several studies have resulted in a better outcome of patients' therapy, especially in patients who need long-term adherence and compliance with drug treatment. It is hypothesized that patients' quality of life of HIV-TB co-infection patients will be improved with the intervention conducted by the pharmacist.

Objective:

In general, the study aimed to evaluate the utility of study participants with specific aims to describe the number of DRP and interventions applied, to describe drug concentration in selected participants (TB drugs: Rifampicin and Pyrazinamide), to compare changes of CD4+ cell counts and plasma HIV RNA (viral load) between baseline and after of intervention, to assess participants compliance and persistence to medication therapy, and descriptive analysis on the direct and indirect costs.

Study design:

This is a prospective, cluster-randomized study with a stepped-wedge design. Clusters correspond to participating centers. A randomly selected center is crossed-over into the intervention with calculation after the start of inclusions within 6-months follow-up in 3 different clinics in Indonesia (Bekasi City Public Hospital, Persahabatan Public Hospital Jakarta and Cipto Mangunkusumo general hospital).

Intervention:

Interventions are given by a pharmacist as a drug consultant is an intervention concerning the drug treatment of HAART and anti-TB. Monthly, patients will have a discussion regarding their medication and drug-related problems they experience. The pharmacist will identify drug-related problems before and during treatment and solve the problems.

Main study parameters/endpoints: change from baseline utility (quality of life) at 6 months Secondary endpoints: changes from baseline in CD4+, VL, adherence, persistence at 6 months and total costs.

DETAILED DESCRIPTION:
1. STUDY BACKGROUND

   1.1 HIV and TB Diseases Human Immunodeficiency Virus (HIV) is a global health concern which the World Health Organization (WHO) estimates that 36.7 million people are living with HIV (PLHIV) with 1.1 million deaths of PLHIV in 2015, worldwide. Among them, there were 2.1 [1.8-2.4] million new HIV infections. Because of its immunosuppressive action, people living with HIV (PLHIV) are prone to be infected with opportunistic infections, such as tuberculosis (TB), pneumonia, and toxoplasmosis. TB itself is known as one of the main risks of death in PLHIV as it considerably accelerates the progression of HIV to AIDS by not only activating viral replication but also accentuating the decline in CD4 cell counts. It is also estimated that TB would affect one-third of the world's population and 9 million new cases of TB are discovered worldwide each year, with more than 1 million cases occurring in patients with HIV or AIDS. The incidence of TB globally has risen enormously since 1990, particularly in certain countries where there is a significant overlap between HIV and TB epidemics. The risk of developing TB is 29 (26-31) times higher in PLHIV than people without HIV as Mycobacterium tuberculosis and HIV are potentiating one another in accelerating the decrease of the immunological function and causing early death.

   HIV treatments have been implemented since the first production of antiretroviral drugs and have been developing fast since because of the increasing number of HIV cases worldwide. The introduction of ARV reduces the development of TB, but this disease continues to occur among PLHIV. Antiretroviral and anti-TB drugs have their complex regimens, and the combination of these drugs in HIV-TB co-infection patients has caused increasingly even more complex regimens, potential toxicities, and issues of adherence due to potential interaction between antiretroviral and anti-TB medications. In HIV patients receiving regular antiretroviral drugs and becoming infected with TB, considerations on the alteration or discontinuation of antiretroviral drugs and selection of TB agents are based upon the efficacy of each selected drug, drug interactions, drug resistance, prevention of treatment failure, and patient adherence.

   1.1.2 Pharmaceutical Care Interventions Such concerning and life-threatening diseases treatments have been massively conducted with a significant success worldwide, marked with the lower incidence of new cases of HIV and TB. However, the major diagnostic and therapeutic deficiencies remain. Health professionals, such as physicians, nurses, pharmacists, and other health professionals are required to ensure the success of HIV TB co-infection therapy based on the guidelines made by international organizations and local governments.

   In the past few decades, there has been a shifting perspective of the pharmacist's role from the traditional role of dispensing medication to the patient-oriented perspective in collaboration with or without other health providers to achieve improvement of patient outcomes as well as the improvement of quality of life. The Pharmaceutical Care (PC) program which involves the specific role of a pharmacist has been implemented mostly in high-income countries to hospitalized- and out-patients. Several systematic reviews and meta-analysis are conducted to evaluate the impact of the patients-oriented intervention in any disease states;8-12 thus the thoroughly and rigorous reviews enable other researchers or health providers to assess and implement the most valid processes of pharmacist intervention in their setting.

   1.1.3 Therapeutic Drug Monitoring in TB Drugs TDM is a multi-disciplinary clinical approach of evaluating and monitoring drug concentration in the blood, defined as the clinical laboratory measurement with proper medical interpretation. It is generally aimed to improve the quality of patient care by adjusting a patient's drug dosage individually within a therapeutic range. A combination of pharmaceutical, pharmacokinetics, pharmacodynamics knowledge and skills are needed to assess the efficacy and safety of particular drugs to achieve a maximum benefit of the patient's drug therapy.

   By far, TDM has been used in many indications, such as to evaluate drug-drug interactions, to assess drug efficacy and safety (toxicity level), and adherence or compliance. However, TDM is not necessarily carried out for all medications. There are several patients' criteria that may have the advantage of TDM, such as: patients with low response of drug treatment that may lead to treatment failure, patients with poor compliance to the treatment, and patients who get treated with narrow therapeutic range drugs (theophylline, aminoglycoside antibiotic, cyclosporine, and lithium). It is believed that TDM has a role in improving TB treatment, especially in TB patients with a low response to the treatment and in HIV/TB co-infection patients. Several studies have conducted TDM and revealed that it could be used as a useful strategy to identify the cause of slow response in TB treatment; thus, it may shorten the time to respond and achieve treatment completion and also optimize ARV dosage when combined with TB drugs.

   1.1.4 Pharmacoeconomics of the pharmacists' interventions There has been an increase in the number of diseases burden worldwide during the past few years which inevitably adding the burden of healthcare expenditures. Many strategies in healthcare settings intended to constrain the expenses, especially to restrict the expenses on drugs. Several studies try to assess the further impact of the intervention from the economic perspective point of view whereas pharmacists as the focus or in a multidisciplinary team. From a public health point of view, pharmacists may actively be involved in health promotion, such as smoking cessation, prevention and treatment of chronic and infectious diseases (e.g., diabetes, hypertension, HIV/AIDS and tuberculosis (TB).
2. STUDY OBJECTIVES

This study aims to evaluate the change in utility (quality of life) of study participants. The specific aims of this study are:

1. To compare the changes of CD4+ cell-counts between baseline and after the study;
2. To compare the difference of plasma HIV RNA (viral load) between baseline and after the study;
3. To assess participants' adherence or compliance to medication therapy (antiretroviral and anti-TB drugs);
4. To assess the direct costs and indirect costs of the pharmacists' interventions.

3. STUDY DESIGN AND SETTING

3.1 STUDY DESIGN

The HIV-TB IND02017 study is a prospective, stepped wedge cluster randomized trial where stepwise randomization occurs at a clinic level. Clinics will be randomized to one of three roll-out schedules, each contributing at least one-month control period and one-month intervention period to the analysis. Data will be collected at the level of the individual, even though the randomization will be implemented at a clinic level. A stepped wedge design (SWD) is a type of crossover design in which different clusters will receive both control and intervention activities with varying points of time. It usually starts with all clusters in the control period, and at subsequent time points, each cluster will receive the intervention period with different duration of the intervention period. This design is being acknowledged in recent years for pragmatic reasons, such as in the HIV disease where there is a strong belief that adding new intervention will give good results than harms for patients with a higher risk of ethical issues if they are randomized into control and intervention groups. SWD has advantages compared to a parallel and crossover design, whereas SWD only needs fewer clusters and samples, useful in trial with resources and cost constraints and ethically acceptable since all the participants in clusters will receive the interventions.

3.2 STUDY SETTING

The study of the impact of pharmacist intervention on improvement of quality of life of TB-infected HIV patients will be implemented in 3 hospital clinics in Jakarta and West Java (Bekasi public hospital, Persahabatan public hospital, and Cipto Mangunkusumo General Hospital Jakarta). The intervention program across each of these sites is 6-months in length or until treatment completion and will be operated in community clinics as this study has targeted HIV/TB outpatients. Pharmacists are the investigators in this study. Participants will be followed for their medication therapy and evaluated by the investigator during the study with the monthly intervention and counseling session at the time of medicine pick up.

4. STUDY POPULATION

4.1 POPULATION

The study will include all HIV patients who develop TB disease at the time of the study at three participating hospital sites, and the follow-up patients will also be applied and maintained throughout the study. Identification of TB disease classification in HIV patients is based on the WHO standard guidelines for tuberculosis and Pedoman Nasional Pengendalian Tuberculosis 2014 (the 2014 Tuberculosis Control National Guidelines), which will include smear sputum results, chest X-ray, and geneXpert (if applicable).

4.2 INCLUSION AND EXCLUSION CRITERIA Will be elaborated in the next section.

4.3 SAMPLE SIZE CALCULATION

The sample size calculation for the stepped wedge design is based on Hemming et al.48 We considered a small effect size of 0.30 with the statistical power of 80% and 5% significance in this study because no studies were investigating the effect of pharmacist intervention in HIV-TB co-infection patients. Based on the assumption and t-test calculation on individual randomization, such design would need 352 study participants (176 per arm). An intra-cluster correlation (ICC) of 0.05 is assumed with the meaning of little correlation between the clusters, which leads to a design effect of 2.12 in the stepped wedge model. With a fixed number of 3 clusters (k), time of observation (t) of 5, the number of observations (m) of 2, and 20% losses of follow-up patients, the sample size is calculated by N = 92 patients.

Calculations of the sample size of stepped wedge model are as follows:

Design effect (DE-SW) Formula:

Total sample size per cluster : M = m x (t+1) = 2 x (5+1) = 12 participants Total study sample size : N = M x k = 12 x 3 = 36 participants Total required sample size : N = N x DE = 36 x 2.12 = 76.32 participants Total sample size : N = 76.32 + 20% excess ≈ 92 participants (anticipated)

Notations:

m : the number of observations made in each cluster: 2 = quality of life and adherence/monitoring drug therapy; k : the number of clusters: 3 clusters (a fixed number of clusters) t : the number of steps: 5 (5 months) t+1 : the number of time points of study implementation (6 time points: before starting the study (time point 1), after month 1 (time point 2), after month 2 (time point 3), etc.)

5. MEASUREMENTS

Measurements included in the study are:

1. Drug-Related Problem (DRP);
2. The number of interventions;
3. TB outcome;
4. Adherence;
5. Persistence;
6. Quality of life;

8) Direct costs; 9) Indirect costs.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 18 years or older;
2. diagnosed with the HIV disease and co-infected with the definite TB disease (PTB or EPTB) during the study period, proven by geneXpert (if applicable), positive smear sputum, and chest X-ray;
3. definite TB patients who are found infected with HIV;
4. attending for outpatient care;
5. can read and write in Indonesian language;
6. not pregnant;
7. taking ARV/HAART at the time of research and is just about to start TB treatment and receive first line of TB drugs;
8. taking ARV/HAART at the time of research and in TB treatment until maximum 3 months from the first consumption of TB drugs and receive first line of TB drugs;
9. HIV patients on TB therapy but have not received ARV/HAART yet;
10. and patients who are willing to take part in this study (signing the informed consent).

Exclusion Criteria:

1. Patients who are diagnosed with only the HIV disease or with other non-TB diseases as reported in their medical records, such as hepatitis C;
2. patients who have enrolled in another clinical trial that may change the nature of basic treatment;
3. patients with limited clinical condition due to their severe condition and therefore are not able to attend outpatient visit, such as stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Monthly evaluation on the participants' quality of life (utility) using the EQ5D-5L questionanire between groups | baseline, 1,2,3,4,5, and 6 months
  To compare the differences in the utility score between the intervention group and control group every study month for 6 months. Utility will be evaluated into 2 scores, i.e utility score (score range: 0-1) and visual analog scale (score range: 0-100). The higher the score the better the utility

SECONDARY OUTCOMES:
Comparison of difference in CD4 cell counts between groups | Baseline and 6 months
  To compare the mean of difference in CD4 cell counts between groups at baseline and after 6 months
Comparison of difference in plasma HIV RNA (viral load) between groups | Baseline and 6 months
  To compare the mean of difference in plasma viral load between groups at baseline and after 6 months
Comparison of difference in participants' medication adherence between groups | Baseline and 6 months
  To compare the mean of difference in the adherence between groups at baseline and after 6 months. Monthly evaluation of medication adherence is measured by pills counting.
Comparison of difference in participants' persistence to attend the study sessions between groups | Baseline and 6 months
  To compare the mean of difference in the persistence between groups at baseline and after 6 months. Monthly evaluation of patient persistence is measured by participant's attendance to the clinic to consult the pharmacist (as the investigator).

CONTACTS AND LOCATIONS:
Overall Officials: Lusiana R Idrus, Master, Principal Investigator — University of Groningen
Locations (3):
- Indonesia (3):
  - Persahabatan public hospital, Jakarta, Jakarta Timur
  - Bekasi city hospital, Bekasi, West Java
  - Ciptomangunkusumo public hospital, Jakarta Pusat

IPD SHARING:
Plan to Share IPD: Yes
Individual participants data will be available for investigators and limited for collaborators
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: September 2019
Access Criteria: Full data only available for investigators